# Acupuncture Treatment for Individuals with Myasthenia Gravis

**Protocol Number: Version 7** 

National Clinical Trial (NCT) Identified Number: NCT05230082

Principal Investigator: Amanda A. Herrmann, PhD

Site/Sponsor: HealthPartners Neuroscience Center, HealthPartners Clinic St.
Paul Como, and Healing Response Acupuncture & Functional
Neurology/HealthPartners Institute

**Institutional Review Board Number: A21-197** 

**Funded by: Park Nicollet Foundation** 

Date: September 8<sup>th</sup>, 2023

# **CONFIDENTIALITY STATEMENT**

This document is confidential communication. Acceptance of this document constitutes agreement by the recipient that no unpublished information contained herein will be published or disclosed without prior approval of the Principal Investigator or other participating study leadership and as consistent with the terms of the award.

# **Table of Contents**

| - | -MENT OF COMPLIANCE | |
|---|---|---|
| INVES | TIGATOR'S SIGNATURE | |
| 1 | PROTOCOL SUMMARY | |
| 1.1 | Synopsis | |
| 1.2 | | |
| 1.3 | Schedule of activities | |
| 2 | INTRODUCTION | |
| 2.1 | , | |
| 2.2 | | |
| | .2.1 Known Potential Risks | |
| 2 | .2.2 Known Potential Benefits | |
| 2 | .2.3 Assessment of Potential Risks and Benefits | |
| 3 | OBJECTIVES AND ENDPOINTS | |
| 4 | STUDY DESIGN | |
| 4.1 | 5 | |
| 4.2 | , 3 | |
| 4.3 | | |
| 4.4 | , | |
| 5 | STUDY POPULATION | |
| 5.1 | | |
| 5.2 | | |
| 5.3 | Lifestyle Considerations | |
| 5.4 | | |
| 5.5 | Strategies for Recruitment and Retention | |
| 6 | STUDY INTERVENTION(S) OR EXPERIMENTAL MANIPULATION(S) | |
| 6.1 | , | |
| | Study Intervention or Experimental Manipulation Description | |
| | Administration and/or Dosing | |
| 6.2 | • | |
| | .2.1 Interventionist Training and Tracking | |
| 6.3 | | |
| 6.4 | , | |
| 6.5 | . , | |
| | .5.1 Rescue Therapy | |
| 7 | STUDY INTERVENTION/EXPERIMENTAL MANIPULATION DISCONTINUATION AND PARTICI | |
| 7.1 | ONTINUATION/WITHDRAWALDiscontinuation of Study Intervention/Experimental Manipulation | |
| 7.2 | , | |
| 7.3 | Lost to Follow-Up STUDY ASSESSMENTS AND PROCEDURES | |
| 8 8.1 | Endpoint and Other Non-Safety Assessments | |
| 8.2 | • | |
| 0.2 | Jaiety Assessificitis | 10 |

| 8.3 | Adverse Events and Serious Adverse Events | 16 |
|---------|--------------------------------------------------------------|----|
| 8.3.1 | Definition of Adverse Events | 16 |
| 8.3.2 | Definition of Serious Adverse Events | 16 |
| 8.3.3 | Classification of an Adverse Event | 17 |
| 8.3.4 | Time Period and Frequency for Event Assessment and Follow-Up | 18 |
| 8.3.5 | Adverse Event Reporting | 18 |
| 8.3.6 | Serious Adverse Event Reporting | 18 |
| 8.3.7 | Reporting Events to Participants | 19 |
| 8.3.8 | Events of Special Interest | 19 |
| 8.3.9 | Reporting of Pregnancy | 19 |
| 8.4 | Unanticipated Problems | 19 |
| 8.4.1 | Definition of Unanticipated Problems | 19 |
| 8.4.2 | Unanticipated Problems Reporting | 20 |
| 8.4.3 | Reporting Unanticipated Problems to Participants | 20 |
| 9 STA | TISTICAL CONSIDERATIONS | 20 |
| 9.1 | Statistical Hypotheses | 20 |
| 9.2 | Sample Size Determination | 20 |
| 9.3 | Populations for Analyses | 21 |
| 9.4 | Statistical Analyses | 21 |
| 9.4.1 | General Approach | 21 |
| 9.4.2 | Analysis of the Primary Endpoint(s) | 22 |
| 9.4.3 | Analysis of the Secondary Endpoint(s) | 22 |
| 9.4.4 | Safety Analyses | 22 |
| 9.4.5 | Baseline Descriptive Statistics | 22 |
| 9.4.6 | Planned Interim Analyses | 23 |
| 9.4.7 | Sub-Group Analyses | 23 |
| 9.4.8 | Tabulation of Individual Participant Data | 23 |
| 9.4.9 | Exploratory Analyses | 23 |
| 10 SUP | PORTING DOCUMENTATION AND OPERATIONAL CONSIDERATIONS | |
| 10.1 | Regulatory, Ethical, and Study Oversight Considerations | |
| 10.1.1 | Informed Consent Process | |
| 10.1.2 | Study Discontinuation and Closure | |
| 10.1.3 | Confidentiality and Privacy | |
| 10.1.4 | Future Use of Stored Specimens and Data | |
| 10.1.5 | Key Roles and Study Governance | |
| 10.1.6 | Safety Oversight | |
| 10.1.7 | Clinical Monitoring | |
| 10.1.8 | Quality Assurance and Quality Control | |
| 10.1.9 | Data Handling and Record Keeping | |
| 10.1.10 | | |
| 10.1.11 | <b>5</b> , | |
| 10.1.12 | Conflict of Interest Policy | 27 |

| 10.2 | Additional Considerations27 |
|------|-----------------------------------|
| 10.3 | Abbreviations and Special Terms27 |
| 10.4 | Protocol Amendment History29 |
| 11 | REFERENCES30 |

# STATEMENT OF COMPLIANCE

The trial will be carried out in accordance with International Council on Harmonisation Good Clinical Practice (ICH GCP) and the following:

• United States (US) Code of Federal Regulations (CFR) applicable to clinical studies (45 CFR Part 46, 21 CFR Part 50, 21 CFR Part 56, 21 CFR Part 312, and/or 21 CFR Part 812).

Investigators and clinical trial site staff who are responsible for the conduct, management, or oversight of clinical trials have completed Human Subjects Protection and ICH GCP Training.

The protocol, informed consent form(s), recruitment materials, and participant materials will be submitted to the Institutional Review Board (IRB) for review and approval. Approval of both the protocol and the consent form(s) must be obtained before any participant is consented. Any amendment to the protocol will require review and approval by the IRB before the changes are implemented to the study. All changes to the consent form(s) will be IRB approved; a determination will be made regarding whether a new consent needs to be obtained from participants who provided consent, using a previously approved consent form.

# **INVESTIGATOR'S SIGNATURE**

The signature below constitutes the approval of this protocol and provides the necessary assurances that this study will be conducted according to all stipulations of the protocol, including all statements regarding confidentiality, and according to local legal and regulatory requirements and applicable US federal regulations and ICH guidelines, as described in the *Statement of Compliance* above.

Signed: Date:

Name: Amanda A. Herrmann, PhD

Title: Research Associate

Principal Investigator or Clinical Site Investigator:

**Investigator Contact Information** 

Affiliation: HealthPartners Neuroscience Center

Address: 295 Phalen Blvd. St. Paul, MN 55130

Mailstop 41200A

Telephone: (651) 495-6356

Email: Amanda.A.Herrmann@HealthPartners.com

# L PROTOCOL SUMMARY

#### 1.1 SYNOPSIS

Title: Acupuncture Treatment for Individuals with Myasthenia Gravis

IRB Number: A21-197

**Study Description:** The purpose of the study is to determine the effect acupuncture

treatment on individuals with a diagnosis of Myasthenia Gravis (MG). A total of 25 people with MG will be enrolled in this study to receive acupuncture treatment 2 times a week for 12 weeks. Participants will be randomized into two groups: 1) Immediate start and 2) Delayed start (12 weeks). The delayed start group will act as a control group for the first 12 weeks, but then receive acupuncture treatment for 12 weeks. We hypothesize that patients with MG who receive

acupuncture treatment will have improved quality of life and activities

of daily living compared to no treatment.

**Specific Aims:** Specific Aim 1: To determine the effect of acupuncture treatment on

quality of life in individuals with MG.

Specific Aim 2: To determine the effect of acupuncture treatment on

activities of daily living in individuals with MG.

Endpoints: Primary Endpoint: Myasthenia Gravis Quality of Life Scale (MG-QOL15)

Secondary Endpoint: Myasthenia Gravis Activities of Daily Living Scale

(MG ADL).

**Study Population:** 25 individuals aged 18-80 with a diagnosis of MG will be recruited for

this study.

**Description of** 

**Sites/Facilities Enrolling** 

**Participants:** 

For in-person visits, participants will receive acupuncture treatment at HealthPartners Neuroscience Center, HealthPartners Clinic St. Paul Como, or Healing Response Acupuncture & Functional Neurology.

Description of Study

Intervention/Experimental

**Manipulation:** 

Acupuncture treatment will be administered by a licensed

acupuncturist for a duration of 12 weeks. Both groups will receive a

total of 24 treatments.

**Study Duration:** The duration of this study is 2 years.

**Participant Duration:** We anticipate that participants will complete all study-related tasks

within approximately 8 months.

#### 1.2 SCHEMA



# 1.3 SCHEDULE OF ACTIVITIES

| | Pre-<br>screening | Pre-<br>treatment<br>1 | Pre-<br>treatment<br>2 | Study<br>Intervention | Post-<br>treatment<br>1 | Post-<br>treatment<br>2 | 2-week<br>follow<br>up call |
|---|---|---|---|---|---|---|---|
| Group 1:<br>Immediate<br>Start | Visit 0 | Visit 1 | N/A | Visit 2-25 | Visit 26 | Visit 27 | N/A |
| Group 2:<br>Delayed Start | | Visit 1 | Visit 2 | Visit 3-26 | Visit 27 | N/A | Visit 28 |
| Review<br>Eligibility | Х | | | | | | |
| Informed<br>Consent | | Х | | | | | |
| Randomization | | Х | | | | | |
| Demographics | | Х | | | | | |
| Medication<br>Review | | Х | х | Х | х | Х | |
| Symptom<br>Severity Scale<br>(Treatment Log) | | | | Х | х | х | Х |
| MG-QOL15 | | Х | Х | | Х | Х | |
| MG-ADL | | Х | Х | | Х | Х | |
| Adverse Events<br>(AE) Reporting | | | | х | х | Х | Х |
| Treatment<br>Adherence | | | | Х | | | |

# **VISIT SCHEDULE DESCRIPTION**

All in-person visits will take place at: HealthPartners Neuroscience Center, 295 Phalen Boulevard, St. Paul, MN, 55130, HealthPartners Clinic St. Paul Como, 2500 Como Ave, St. Paul, MN 55108, or Healing Response Acupuncture & Functional Neurology, 11550 Stillwater Blvd N. Suite 101, Lake Elmo, MN 55402.

# 1. Pre-screening Phone Call (Groups 1 & 2)

- <u>Duration:</u> Approximately 30 minutes
- Research staff will:
  - Provide potential participants information about the study and ask whether they are interested in participating.
  - o Determine whether they meet the inclusion/exclusion criteria for the study.
  - o Ask participants for permission to communicate through e-mail for the study
  - o Assist participants with setting up an e-mail account, if they do not have one.

 Schedule Pre-treatment Visit if the person is eligible for the study and e-mail the person the Informed Consent, Health Insurance Portability and Accountability Act (HIPPA), and HealthPartners non-discrimination forms.

# 2. Pre-treatment Visit 1 (Groups 1 & 2)

- <u>Duration:</u> Approximately 1 hour via phone
- Research staff will:
  - o Review the Informed Consent and HIPPA documents with potential participants.
  - Answer any questions of potential participants and ensure they understand the expectations of the study.
  - Ask participants to electronically sign the Informed Consent and HIPAA documents via Research Electronic Data Capture (REDCap), a secure web-based system, and provide them electronic copies for their records.
  - Complete the Demographics and Medication Review short forms in the relevant electronic case report forms (eCRFs) in REDCap.
  - Interview patients using the Myasthenia Gravis Quality of Life Scale (MG-QOL15) and Activities of Daily Living (MG ADL) surveys and document in REDCap.

# 3. Pre-treatment Visit 2 (Group 2 only)

- Duration: Approximately 20 minutes via phone
- Research staff will:
  - Complete the Medication Review short form in the relevant electronic case report forms (eCRFs) in Research Electronic Data Capture (REDCap), a secure web-based system.
  - Interview patients using the MG-QOL15 and MG ADL surveys and document in REDCap.

# 4. Study Intervention (Groups 1 & 2)

- Duration: Each visit approximately 1 hour
- A study acupuncturist will:
  - Complete the Adverse Events (AE) Reporting, Medication Review, and Treatment Adherence in the relevant eCRFs in REDCap.
  - o Perform the acupuncture treatment.

# 5. Post-treatment Visit 1 (Groups 1 & 2)

- <u>Duration:</u> Approximately 20 minutes via phone
- Research staff will:
  - Complete the AE Reporting and Medication Review forms in the relevant eCRFs in REDCap.
  - Interview patients using the Symptom Severity Scale (from the treatment log),
     MG-QOL15, and MG ADL surveys and document in REDCap.
  - Ask qualitative survey questions about the participant's experience with acupuncture.

# 6. Post-treatment Visit 2 (Group 1 only)

- Duration: Approximately 20 minutes via phone
- Research staff will:

- Complete the AE Reporting and Medication Review forms in the relevant eCRFs in REDCap.
- Interview patients using the Symptom Severity Scale (from the treatment log),
   MG-QOL15, and MG ADL surveys and document in REDCap.
- Ask qualitative survey questions about the participant's experience with acupuncture.

# 7. 2-week follow up call (Group 2 only)

- <u>Duration</u>: Approximately 5 minutes via phone
- Research staff will:
  - o Complete the AE Reporting in the relevant eCRFs in REDCap.
- 8. Early Withdrawal Call (for individuals who withdraw from the study early)
  - <u>Duration:</u> Approximately 20 minutes via phone
  - Research staff will:
    - Complete the AE Reporting and Medication Review forms in the relevant eCRFs in REDCap.
    - Interview patients using the Symptom Severity Scale (from the treatment log), MG-QOL15, and MG ADL surveys and document in REDCap.Ask qualitative survey questions about the participant's experience with acupuncture.

#### 2 INTRODUCTION

# 2.1 BACKGROUND & STUDY RATIONALE

Myasthenia gravis (MG) is an autoimmune disease in which antibodies bind to acetylcholine receptors or at the neuromuscular junction, causing muscle weakness.<sup>1</sup> It is a rare disease affecting approximately 8-10 people per 1 million people each year.<sup>2</sup> Weakness is typically more proximal than distal and can be generalized or localized.<sup>1</sup> Common symptoms are muscle weakness, fatigue, ptosis, and diplopia. Symptoms can also include impaired speaking, swallowing, and chewing. MG can typically be managed well through medication therapy, including cholinesterase inhibitors, corticosteroids, and immunosuppressants. However, in a recent systematic review, acupuncture was shown to have a significant positive effect in treating MG and might enhance the efficacy of medications.<sup>3</sup>

Acupuncture is a non-pharmacologic treatment that has been practiced in Chinese medicine for over 4,000 years.<sup>4</sup> It is a technique where fine needles are inserted into specific areas of the body to achieve a therapeutic benefit.<sup>4</sup> Historically, acupuncture is based on a Chinese/East Asian medical theory that acupuncture restores normal function to the body by balancing Qi.<sup>4</sup> Acupuncture has been used and reported by physicians in the United States as early as the 1600s and has been researched since the 1800s. Most of the early reports were of individual patient cases, whereas the first randomized controlled trial of acupuncture treatment was published in 1975. Acupuncture has been shown to be safe and effective treatment for treating several chronic conditions, including patients suffering from headache,<sup>5</sup> migraine,<sup>5</sup> and chronic pain.<sup>6</sup> Although both minor and serious adverse events (AEs) have been reported, serious complications related to acupuncture are rare.<sup>7</sup>

A recent systematic review and meta-analysis done by Zhang and colleagues examined 13 randomized controlled trials, which included 775 people with MG that were treated with acupuncture.<sup>3</sup> The primary outcome measure was the relative clinical score response rate, which is the primary assessment that is used to evaluate the severity and treatment effect of MG in China.<sup>8</sup> The review concluded that integrative long-term therapy, including acupuncture and medication, may be helpful for individuals with MG.<sup>3</sup> However, the authors also concluded that more rigorous studies and longer follow-up times are needed.<sup>3</sup> Thus, the primary goal of this study is to examine the effect of acupuncture on quality of life and the activities of daily living in patients with MG.

# 2.2 RISK/BENEFIT ASSESSMENT

#### 2.2.1 KNOWN POTENTIAL RISKS

# **Acupuncture Treatment**

Reported Side Effects<sup>9</sup>:

| Common | Uncommon | Rare | Very Rare |
|---|---|---|---|
| 1-10 out of 100 people | 1-10 out of 1,000 people | 1-10 out of 10,000 people | <1 out of 10,000 people |
| Bleeding | Inflammation/swelling | Local infection | Palpitations |
| Hematoma (bleeding outside of vessels) | Bruising | Redness | Constipation |
| | Pain during needling | Itching | Diarrhea |
| | Local muscle pain | Sweating | Gastrospasm<br>(stomach spasm) |
| | Nerve irritation or injury | Decrease/increase of blood pressure | Enterospasm (spasm of the intestine) |
| | Headache | Unconsciousness | Weight loss |
| | Fatigue | Tachycardia | Circulatory disturbance |
| | Dizziness | Breathing difficulties | Lesion of blood vessels |
| | Nausea | Vomiting | Systemic infection |
| | Exacerbation of symptoms that led to treatment | Worsening health state | Euphoria |
| | | Generalized muscle pain | Nightmares |
| | | Restricted movement | Poor concentration |
| | | Joint problems | Imbalance |
| | | Feeling of coldness | Disturbance of speech |
| | | Menstrual problems | Disorientation |
| | | Depressive mood | Shivering |
| | | Anxiety | Eye irritation |
| | | Sleep disturbance | Broken (retained)<br>needles |
| | | Restlessness/nervousness | Organ puncture/ Pneumothorax |
| | | Disturbed vision | Injury of the central nervous system |

| Tinnitus | Injury of the |
|----------|---------------|
| Tinnitus | pericardium |

# Assessments/Questionnaires (MG-QOL15 & MG ADL)

The Myasthenia Gravis Quality of Life Scale short form self-assessment (MG-QOL15) and Activities of Daily Living self-assessment (MG ADL) are standardized questionnaires that will measure personal perception of life and activities of daily living. The questions on these assessments may make participants feel uncomfortable because some parts may be easy to answer, while some parts may be difficult or tiring. Filling out the questionnaires may also cause individuals to feel uncomfortable or upset.

# **Loss of Confidentiality**

There may be a slight possibility of breach of confidential information that was collected. However, the following procedures will be implemented to reduce this risk:

- Data collection and reporting tools will be developed and stored internally.
- Data collected and stored electronically will remain confidential and secure (e.g. secured server and password protected files [REDCap]).
- Study binders will be stored in a locked file cabinet within a locked office.
- After the study is closed, all subject identifiers will be destroyed.

#### 2.2.2 KNOWN POTENTIAL BENEFITS

Acupuncture has been shown to be a safe and effective treatment for several patient populations. Although there is less evidence for individuals with MG, acupuncture treatment may improve quality of life and activities of daily living.

# 2.2.3 ASSESSMENT OF POTENTIAL RISKS AND BENEFITS

We believe the potential risks to the participants in this study are minimal and that the benefit of understanding whether acupuncture treatment improves quality of life and activities of daily living in patients with MG outweighs the potential risks.

# **3 OBJECTIVES AND ENDPOINTS**

| OBJECTIVES | ENDPOINTS |
|---|---|
| Primary | |
| To determine the effect of acupuncture on quality of life in patients with MG. | MG-QOL15 |
| Secondary | |
| To determine the effect of acupuncture on activities of daily living in patients with MG. | MG ADL |

#### 4 STUDY DESIGN

#### 4.1 OVERALL DESIGN

# Study Design:

This study is an unblinded, controlled randomized, 2-arm clinical trial.

# **Hypotheses:**

**Primary Hypothesis:** We hypothesize that acupuncture will improve the quality of life in MG patients. **Secondary Hypothesis:** We hypothesize that acupuncture will improve activities of daily living in MG patients.

#### Randomization:

Prior to the first acupuncture treatment visit, participants will be randomized into two treatment groups. Randomization is explained in **Section 6.3**.

# Acupuncture Treatment Groups:

**Group 1:** 10 participants will receive acupuncture treatment immediately 2x per week for 12 weeks = 24 total.

**Group 2:** After a 12-week delay, 10 participants will receive acupuncture treatment 2x per week for 12 weeks = 24 total.

# Study Intervention:

Acupuncture treatment will consist of a standardized treatment protocol designed for this study. Approximately 23-32 needles will be inserted into specific areas of the body for a duration of 30 minutes. Additional details of the treatment are discussed in **Section 6.1**.

#### 4.2 SCIENTIFIC RATIONALE FOR STUDY DESIGN

<u>Justification for an unblinded study:</u> Because it will be clear to both study personnel and participants who will have a delayed start and who will start immediately, neither will be blinded in this study. This will be reported as a limitation of the study.

Justification for an uncontrolled study with no control group: N/A

#### 4.3 JUSTIFICATION FOR INTERVENTION

Acupuncture is a treatment that has been practiced for over 4,000 years and is well-accepted by many cultures. Although the mechanism is not well understood, acupuncture has been shown to be safe and effective for treating several conditions (e.g. headaches, chronic pain). The purpose of this study is to determine whether acupuncture treatment can improve quality of life and activities of daily living in patients with MG.

#### 4.4 END-OF-STUDY DEFINITION

A participant is considered to have completed the study if he or she has completed study treatment visits and assessments. The end of the study is defined as completion of the last post-treatment visit for each group.

# STUDY POPULATION

#### 5.1 INCLUSION CRITERIA

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

- Ability to provide and provision of signed and dated informed consent form
- Age 18-80
- · Diagnosis of MG

#### 5.2 EXCLUSION CRITERIA

An individual who meets any of the following criteria will be excluded from participation in this study:

- Non-English speaking
- Participation in acupuncture treatment outside of the study, while enrolled
- History of any other serious neurological, psychiatric, chronic pain disorders, or seizures
- History of bleeding diathesis, other bleeding disorders, or syncope with needle puncture
- Recent or active substance use disorder
- Women who are currently pregnant, lactating, or planning to become pregnant during the study
- Any other medical conditions that could affect their ability to participate in acupuncture treatments for the study duration (as determined by study investigators)
- Active participation or past participation ≤3 months in any other interventional study.
- Unwilling to participate in all study related activities

# 5.3 LIFESTYLE CONSIDERATIONS

N/A

# 5.4 SCREEN FAILURES

#### **Pre-screening Phone Call:**

All potential participants will undergo a pre-screening phone call to determine whether they meet the inclusion/exclusion criteria. Patients will be considered <u>ineligible</u> if they do not meet one or more of the inclusion/exclusion criteria during pre-screening. We will collect information on why participants are ineligible or decide not to move forward with the trial.

#### **Pre-treatment Visit:**

<u>Screen failures</u> are defined as participants who are considered eligible during the pre-screening phone call, but it was subsequently determined that they do not meet one or more of the inclusion/exclusion criteria at or after the Pre-treatment (baseline) visit. We will collect information on why participants screen fail or decide not to move forward with the trial.

# **Rescreening Patients:**

Individuals who do not meet the criteria for participation in this trial (ineligible or screen failure) because of meeting one or more exclusion criteria that are likely to change over time may be rescreened up to one time. Examples include: successful treatment for a substance use disorder; women who are no longer

pregnant, lactating, or planning to become pregnant; or participation in an interventional study ≥3 months prior. Rescreened participants will be assigned a new participant number.

#### 5.5 STRATEGIES FOR RECRUITMENT AND RETENTION

**Recruitment:** Individuals with MG will be recruited by physician and therapist referrals from HealthPartners' clinics. We will also advertise our research study by distributing flyers to HealthPartners' physicians and throughout HealthPartners' clinics. Recruitment flyers will also be provided to our community partners for example, the Minnesota Brain Injury Alliance, TRIA, and Allina Health. If we encounter difficulties with recruitment, we plan to submit an amendment to the IRB to contact HealthPartners and Park Nicollet patients and members and invite them to participate.

To reach our target enrollment, we anticipate that we will need to screen 60 people, of those 30 individuals will sign the informed consent, and of those 25 individuals will be randomized to treatment groups.

**Remuneration:** Participants will be provided gift cards totaling \$50 per person for completing certain time points of the research study. Group 1: Will receive a \$25 gift card after all acupuncture treatments and surveys were completed, and another \$25 gift card after the last post treatment visit, if all surveys were completed. Group 2: Will receive a \$25 gift card after half of the acupuncture treatments have been completed and surveys were completed, and another \$25 after the post-treatment visit, if all surveys were completed.

# 6 STUDY INTERVENTION(S) OR EXPERIMENTAL MANIPULATION(S)

#### 6.1 STUDY INTERVENTION(S) OR EXPERIMENTAL MANIPULATION(S) ADMINISTRATION

# 6.1.1 STUDY INTERVENTION OR EXPERIMENTAL MANIPULATION DESCRIPTION

The study intervention for both groups is acupuncture treatment. Acupuncture is a treatment where fine needles are inserted into specific areas of the body to achieve a therapeutic benefit. The treatment regimen is described next in more detail.

#### 6.1.2 ADMINISTRATION AND/OR DOSING

# **Acupuncture Treatment Methods:**

Group 1 will receive twice-weekly acupuncture immediately over 12-weeks. After a 12-week delay, Group 2 will also receive twice-weekly acupuncture over 12-weeks. Acupuncture treatments will be separated by a minimum of 2 days and a maximum of 14 days, unless a participant has an illness, such as COVID-19. In this case, additional time may be allowed, as determined by the investigator. Treatment methods will be identical for both groups and are described below.

Standard, sterile stainless-steel, disposable needles (DongBang™ Corporation, Spring Ten 0.22 x 30mm; Boryeoung, Republic of Korea) will be inserted in the acupuncture point locations (described below), with approximately 23-32 needles used for each treatment session. The number of needles used will be based

on the patient-reported symptoms. The depth of the needle insertion will be approximately 10-20mm, depending on the region of the body undergoing treatment. Needle reaction (soreness, numbness or distended feeling around the point, also known as a Deqi sensation) will occur during the initial insertion. Following 10 minutes of retention, some of the needles will be rotated in order to maintain Deqi sensation. Maintaining Deqi sensation has been shown to increase the effectiveness of acupuncture. All needles will be left in place for a total of 30 minutes, which is a typical duration in acupuncture practice.

Acupuncture points were selected for their classical Traditional Chinese Medicine indications relevant to MG symptom pathology, as well as their modern biomedical muscular, immunological, and neurological actions. The anatomical location for each point will be based on the World Health Organization's acupuncture point guideline.<sup>12</sup> Traditional Chinese manual acupuncture will be used at up to 32 acupuncture points. During treatment, acupuncture needles can be removed due to extreme pain or discomfort, so as not to exceed the removal of more than 4 needles.

#### 6.2 FIDELITY

### 6.2.1 INTERVENTIONIST TRAINING AND TRACKING

#### **Acupuncturists:**

Acupuncture treatments will be administered by MN licensed acupuncturists with a Master's degree level of training in acupuncture (or higher) from accredited institutions, and five or more years of clinical experience. Prior to enrolling participants, the acupuncturists will complete practice sessions together of the treatment protocol and methods of administration to ensure consistency between providers.

# Training:

Following IRB approval and prior to recruitment and enrollment, the study acupuncturists will complete at least 1 practice session each. For the training, we will seek volunteers who will sign a volunteer consent form prior to participating. The purpose of training will be to ensure consistency in intervention procedures and further standardized treatment methods. This includes, but is not limited to: needle location, needle depth, time of first and last needle placement, and total treatment duration.

#### Tracking:

All practice sessions will be documented on a training log. This will include dates and times of the trainings, names of the volunteers, and printed names and signatures of the study acupuncturists. We will also keep a record of the volunteers' signed treatment release forms.

# 6.3 MEASURES TO MINIMIZE BIAS: RANDOMIZATION AND BLINDING

#### Randomization:

Randomization will be performed with a 1:1 allocation ratio. Balanced treatment assignments will be achieved using permuted block randomization with random block sizes stratified by gender. This decision was based on evidence that females in this population reported higher rates of headaches.<sup>13</sup> The study biostatistician will generate a randomization schedule using the SURVERYSELECT procedure in SAS. Assignments will not be seen by other study personnel in advance and will not be changed after randomization.

# Blinding:

Study personnel will be unblinded to the randomization, as it will be clear the number of participants who have a 12-week delay and those who do not. In addition, it will be clear to participants which treatment group they are in and it will be impossible to blind them from this information.

#### 6.4 STUDY INTERVENTION/EXPERIMENTAL MANIPULATION ADHERENCE

Participants will be asked to adhere to study visits and to complete study assessments. Participants will remain active unless withdrawn from the study (see **Section 7**). We will track participants' adherence to study visits, as well as completion of the assessments. These will be documented in the relevant eCRF.

#### 6.5 CONCOMITANT THERAPY

For this protocol, participants may use non-opioid analgesics for pain control, including over-the-counter medications and dietary supplements, and prescribed medications. This includes use for rescue therapy in the event of exacerbation of symptoms due to acupuncture treatment. Medication usage will be assessed at each study visit and documented in the relevant eCRF.

#### 6.5.1 RESCUE THERAPY

See section 6.5 (above).

# 7 STUDY INTERVENTION/EXPERIMENTAL MANIPULATION DISCONTINUATION AND PARTICIPANT DISCONTINUATION/WITHDRAWAL

#### 7.1 DISCONTINUATION OF STUDY INTERVENTION/EXPERIMENTAL MANIPULATION

When a participant who signed the consent form chooses to discontinue participation in the study or study intervention, or if the principal investigator and co-investigators determine that a participant should discontinue participation, they will be withdrawn from the study. A withdrawal will either be defined as 'Patient Withdrawal' or 'Principal Investigator Withdrawal'. The participant will be asked to complete an early withdrawal phone call 7-14 days from the date the intervention was discontinued. The purpose of the phone call will be to record any AEs or serious adverse events (SAEs) that may have occurred after the discontinuation of treatment. Research staff will attempt to call the participant up to 3 times.

The data that will be collected at the time of study withdrawal will include the following:

The reason(s) for discontinuation of the study intervention

The data that will be collected during the early withdrawal phone call will include the following:

AEs or SAEs that occurred since the time of withdrawal

# 7.2 PARTICIPANT DISCONTINUATION/WITHDRAWAL FROM THE STUDY

Participants are free to withdraw from participation in the study at any time upon request. An investigator may discontinue a participant from the study for the following reasons:

1. Participant has not completed an acupuncture treatment for > 14 days, unless a participant has an illness, such as COVID-19. In this case, additional time may be allowed, as determined by the investigator.

- 2. Significant study intervention non-compliance
- 3. Lost-to-follow up; unable to contact subject (see Section 7.3, Lost to Follow-Up)
- 4. Any event or medical condition or situation occurs such that continued collection of follow-up study data would not be in the best interest of the participant or might require an additional treatment that would confound the interpretation of the study
- 5. The participant meets an exclusion criterion (either newly developed or not previously recognized) that precludes further study participation

The reason for participant discontinuation or withdrawal from the study will be recorded on the relevant eCRF. Subjects who sign the informed consent form and are randomized but do not receive the study intervention may be replaced. Subjects who sign the informed consent form, and are randomized and receive the study intervention, and subsequently withdraw, or are discontinued from the study, will not be replaced.

#### 7.3 LOST TO FOLLOW-UP

A participant will be considered lost to follow-up if he or she fails to attend any scheduled study visit and study staff are unable to contact the participant after at least 5 attempts, while maintaining the 7 day maximum between visits.

The following actions must be taken if a participant fails to attend any required study visit:

- Study staff will attempt to contact the participant, reschedule the missed visit, counsel the participant on the importance of maintaining the assigned visit schedule and ascertain if the participant wishes to and/or should continue in the study.
- Before a participant is deemed lost to follow-up, the investigator or designee will make every
  effort to regain contact with the participant (where possible, telephone calls or e-mail if no
  answer leave a voicemail on the first and last attempt). These contact attempts will be
  documented.
- Should the participant continue to be unreachable, he or she will be considered to have withdrawn from the study with a primary reason of lost to follow-up.

# 8 STUDY ASSESSMENTS AND PROCEDURES

#### 8.1 ENDPOINT AND OTHER NON-SAFETY ASSESSMENTS

**Demographics:** Demographic information will be collected, including: gender, age, race, ethnicity, language, height, weight, marital status, employment status, date of MG diagnosis, and e-mail address for study contact).

**Medication Review:** At study enrollment, participants' prescription medications will be recorded and tracked for the study duration. Medication data will be used for exploratory purposes.

**Treatment Adherence:** The participant's treatment adherence will be measured to determine tolerability of acupuncture. We will record the number of attended acupuncture sessions. We will also record participants' ability to maintain the acupuncture duration of 30 minutes per session.

**Symptom Severity Scale:** This scale will assess the participant's usual symptoms of MG and the severity of their symptoms. This scale was custom designed for this study.

**Quality of Life:** Participants will be asked to complete the MG-QOL15,<sup>14</sup> a brief 15-item disease specific questionnaire that is designed to assess aspects of quality of life in Myasthenia Gravis. It includes questions regarding quality of life, such as vision, speaking, eating, and activities.

**Activities of Daily Living:** Participants will be asked to complete the MG-ADL, <sup>15</sup> an eight-item patient-reported scale developed to assess MG symptoms and their effects on daily activities. It combines 2 items on daily life activities (ability to brush teeth or comb hair and ability to arise from a chair) with 6 MG symptoms: diplopia, ptosis, chewing, swallowing, voice/speech problems, and respiratory symptoms.

A strong positive correlation between the MG-ADL and the MG-QOL15 (r=0.76, P<0.0001) has been previously demonstrated.<sup>15</sup>

**Qualitative Feedback Survey:** A list of qualitative feedback survey questions will allow for participant's to discuss their experience with acupuncture treatment.

#### 8.2 SAFETY ASSESSMENTS

#### **Assessment of Adverse and Serious Adverse Events:**

AEs and SAEs will be monitored by acupuncturists during acupuncture treatment sessions, and by study staff. The acupuncturists and research staff will immediately notify the Principal Investigator and utilize the eCRF to record any AEs or SAEs. The PI and the study physician will review and categorize all AEs or SAEs and report them accordingly, as discussed below.

# 8.3 ADVERSE EVENTS AND SERIOUS ADVERSE EVENTS

# 8.3.1 DEFINITION OF ADVERSE EVENTS

This protocol uses the definition of AE from 21 CFR 312.32 (a): any untoward medical occurrence associated with the use of an intervention in humans, whether or not considered intervention-related.

# 8.3.2 DEFINITION OF SERIOUS ADVERSE EVENTS

This protocol uses the definition of SAE from 21 CFR 312.32 (a): An AE or suspected adverse reaction is considered "serious" if, in the view of either the investigator or study clinician, it results in any of the following outcomes: Death, a life-threatening AE, inpatient hospitalization or prolongation of existing hospitalization, a persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions, or a congenital anomaly/birth defect. Important medical events that may not result in death, be life-threatening, or require hospitalization may be considered serious when, based upon

appropriate medical judgment, they may jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the outcomes listed in this definition.

#### 8.3.3 CLASSIFICATION OF AN ADVERSE EVENT

# 8.3.3.1 SEVERITY OF EVENT

For AEs not included in the protocol defined grading system, the following guidelines will be used to describe severity.

- 1. **Mild** Events require minimal or no treatment and do not interfere with the participant's daily activities.
- 2. **Moderate** Events result in a low level of inconvenience or concern with the therapeutic measures. Moderate events may cause some interference with functioning.
- 3. **Severe** Events interrupt a participant's usual daily activity and may require systemic drug therapy or other treatment. Severe events are usually potentially life-threatening or incapacitating. Of note, the term "severe" does not necessarily equate to "serious".

# 8.3.3.2 RELATIONSHIP TO STUDY INTERVENTION/EXPERIMENTAL MANIPULATION

All AEs will have their relationship to study procedures, including the intervention, assessed by an appropriately-trained clinician based on temporal relationship and his/her clinical judgment. The degree of certainty about causality will be graded using the categories below.

- Definitely Related There is clear evidence to suggest a causal relationship, and other possible
  contributing factors can be ruled out. The clinical event, including an abnormal laboratory test
  result, occurs in a plausible time relationship to study procedures administration and cannot be
  explained by concurrent disease or other drugs or chemicals. The response to withdrawal of the
  study procedures should be clinically plausible. The event must be pharmacologically or
  phenomenologically definitive.
- Probably Related There is evidence to suggest a causal relationship, and the influence of other
  factors is unlikely. The clinical event, including an abnormal laboratory test result, occurs within a
  reasonable time after administration of the study procedures, is unlikely to be attributed to
  concurrent disease or other drugs or chemicals, and follows a clinically reasonable response on
  withdrawal.
- Potentially Related There is some evidence to suggest a causal relationship (e.g., the event occurred within a reasonable time after administration of study procedures). However, other factors may have contributed to the event (e.g., the participant's clinical condition, other concomitant events). Although an AE may rate only as "possibly related" soon after discovery, it can be flagged as requiring more information and later be upgraded to "probably related" or "definitely related", as appropriate.
- Unlikely to be related A clinical event, including an abnormal laboratory test result, whose temporal relationship to study procedures administration makes a causal relationship improbable (e.g., the event did not occur within a reasonable time after administration of the study procedures) and in which other drugs or chemicals or underlying disease provides plausible explanations (e.g., the participant's clinical condition, other concomitant treatments).

Not Related – The AE is completely independent of study procedures administration, and/or
evidence exists that the event is definitely related to another etiology. There must be an
alternative, definitive etiology documented by the clinician.

# 8.3.3.3 EXPECTEDNESS

A clinician with expertise in MG will be responsible for determining whether an AE is expected or unexpected. An AE will be considered unexpected if the nature, severity, or frequency of the event is not consistent with the risk information previously described for the study procedures.

# 8.3.4 TIME PERIOD AND FREQUENCY FOR EVENT ASSESSMENT AND FOLLOW-UP

The occurrence of an AE or SAE may come to the attention of study personnel during study visits and interviews of a study participant.

All AEs, not otherwise precluded per the protocol, will be captured on the appropriate eCRF. Information to be collected includes event description, time of onset, clinician's assessment of severity, relationship to study procedures (assessed only by those with the training and authority to make a diagnosis), and time of resolution/stabilization of the event. All AEs occurring while on study will be documented appropriately regardless of relationship. All AEs will be followed to adequate resolution.

Any medical or psychiatric condition that is present at the time that the participant is screened will be considered as baseline and not reported as an AE. However, if the study participant's condition deteriorates at any time during the study, it will be recorded as an AE.

Changes in the severity of an AE will be documented to allow an assessment of the duration of the event at each level of severity to be performed. Documentation of onset and duration of each episode will be maintained for AEs characterized as intermittent.

Study staff will record events with start dates occurring any time after the first acupuncture treatment session until the last post-treatment visit for each group. After the first acupuncture study and until study completion, study staff will inquire about the occurrence of AE/SAEs. All reported events will be monitored until the last post-treatment visit for each group. We will also conduct a 2-week follow up phone call for Group 2 to collect information on any advese events. Any reported event that is definitely or probably related to the intervention will be followed until resolution or stabilization.

#### 8.3.5 ADVERSE EVENT REPORTING

In consultation with the Principal Investigator (PI) and the study clinician, a trained member of the study team will be responsible for conducting an evaluation of an AE and shall report the results of such evaluation to the reviewing IRB either at the time of continuing review or within 10 working days of becoming aware of the event if the event is considered to be serious or meets the definition of an unanticipated problem involving risks to study subjects or others.

#### 8.3.6 SERIOUS ADVERSE EVENT REPORTING

In consultation with the PI and the study clinician, a trained member of the study team will be responsible for conducting an evaluation of a SAE and shall report the results of such evaluation to the reviewing IRB as soon as possible, but in no event later than 10 working days after the investigator first learns of the event.

#### 8.3.7 REPORTING EVENTS TO PARTICIPANTS

Following IRB review of any AEs or SAEs, the PI will follow the IRB's recommended actions. This may include, but is not limited to, modifying the informed consent document or process, re-consenting current participants, providing information to past or current participants (e.g. whenever the information may relate to the participant's willingness to continue participants), and modifications to the protocol/research plan.

# 8.3.8 EVENTS OF SPECIAL INTEREST

N/A

#### 8.3.9 REPORTING OF PREGNANCY

Women who are currently pregnant, lactating, or planning to become pregnant during the study are excluded from this study. This is due to the hormonal changes that may alter headache patterns. If any participant who is still undergoing acupuncture treatment expectedly or unexpectedly becomes pregnant while active in the trial, the participant will be withdrawn from the study by the Principal Investigator. The participant will be asked to complete an early withdrawal phone call in 7-14 days from the date the intervention was discontinued for safety follow-up.

If any participant who has completed all acupuncture treatment sessions expectedly or unexpectedly becomes pregnant, the participant may remain in the study until study completion.

#### 8.4 UNANTICIPATED PROBLEMS

# 8.4.1 DEFINITION OF UNANTICIPATED PROBLEMS

This protocol uses the definition of Unanticipated Problems as defined by the Office for Human Research Protections (OHRP). OHRP considers unanticipated problems involving risks to participants or others to include, in general, any incident, experience, or outcome that meets <u>all</u> of the following criteria:

- Unexpected in terms of nature, severity, or frequency given (a) the research procedures that are
  described in the protocol-related documents, such as the IRB-approved research protocol and
  informed consent document; and (b) the characteristics of the participant population being
  studied;
- 2. Related or possibly related to participation in the research ("possibly related" means there is a reasonable possibility that the incident, experience, or outcome may have been caused by the procedures involved in the research); and
- 3. Suggests that the research places participants or others at a greater risk of harm (including physical, psychological, economic, or social harm) than was previously known or recognized.

#### 8.4.2 UNANTICIPATED PROBLEMS REPORTING

The PI will report unanticipated problems (UPs) to the reviewing IRB. The UP report will include the following information:

- Protocol identifying information: protocol title and number, PI's name, and the IRB project number
- A detailed description of the event, incident, experience, or outcome
- An explanation of the basis for determining that the event, incident, experience, or outcome represents an UP
- A description of any changes to the protocol or other corrective actions that have been taken or are proposed in response to the UP

To satisfy the requirement for prompt reporting, UPs will be reported using the following timeline:

• UPs will be reported to the IRB as soon as possible, but no later than 10 working days after the investigator first learns of the event

# 8.4.3 REPORTING UNANTICIPATED PROBLEMS TO PARTICIPANTS

Following IRB review of any unanticipated problems, the PI will follow the IRB's recommended actions. This may include, but is not limited to, modifying the informed consent document or process, reconsenting current participants, providing information to past or current participants (e.g. whenever the information may relate to the participant's willingness to continue participants), and modifications to the protocol/research plan.

# 9 STATISTICAL CONSIDERATIONS

#### 9.1 STATISTICAL HYPOTHESES

#### Primary:

We hypothesize that quality of life, as assessed by MG-QOL15, will improve with acupuncture treatment compared to no acupuncture treatment.

#### Secondary:

We hypothesize that quality of life, as assessed by MG ADL, will improve with acupuncture treatment compared to no acupuncture treatment.

# 9.2 SAMPLE SIZE DETERMINATION

We anticipate enrolling 10 subjects in each study group. The primary analysis is a two-sided two sample t-test comparing the mean change in MG-QOL15 over 12-weeks weeks from a delayed start 2-group design. We hypothesize that Group 1 who received acupuncture treatment will experience a change in QOL over the 12-weeks while Group 2, the untreated control, will not. We will analyze the data such that the opposite could be shown. The null hypothesis is that there will be no difference between treatment

groups. Our sample size of 10 subjects in each group achieves 80% power at a 5% significance level to detect a 1.32 SD difference in mean change in MG-QOL15 between groups (PASS software version 11). No interim analyses are planned. The potential effect on our power if for a range of true effect sizes are displayed in the table below. If our final analysis shows a smaller effect size than 1.32 SD difference, we will include and post-hoc power analysis with the results.

| N | δ/ σ | Power | Alpha |
|----|------|-------|-------|
| 20 | 0.9 | 0.44 | 0.05 |
| 20 | 1.0 | 0.56 | 0.05 |
| 20 | 1.3 | 0.78 | 0.05 |
| 20 | 1.6 | 0.91 | 0.05 |

N = total sample size, 1:1 Randomization to 2 groups;

 $\delta$  = treatment effect (change);

 $\sigma$  = standard deviation.

Based on preliminary estimates, we do not anticipate difficulty recruiting 20 subjects. HealthPartners clinicians see approximately 4 individuals with MG per month at the Neuroscience Center and Park Nicollet Clinics, approximately 50 annually. Therefore, we will need a 40% enrollment rate to reach our recruitment goal in the allotted time frame. In addition, we also plan to recruit and enroll from other HealthPartners clinics and within the community. If we see a 20% reduction in sample size due to dropout, withdrawal, or missing data, our power will be 71% to detect a similar effect size. This, and other possible changes in power due to attrition, are listed in the table below. \*Note: The original sample size estimation was for 20 individuals; however, we wrote the protocol so that we could replace anyone who did not start the intervention. Thus, we are increasing the enrollment target to 25, which is not reflected in the original power analysis.

| N | δ | σ | Power | Alpha |
|----|-----|---|-------|-------|
| 16 | 9.5 | 7 | 0.71 | 0.05 |
| 18 | 9.5 | 7 | 0.77 | 0.05 |
| 20 | 9.5 | 7 | 0.82 | 0.05 |

N = total sample size;  $\delta$  = treatment effect (change);  $\sigma$  = standard deviation.

#### 9.3 POPULATIONS FOR ANALYSES

All analyses will be performed on an intention-to-treat basis. If poor attendance at acupuncture treatments is observed, we will perform a per-protocol analysis as a sensitivity analysis.

# 9.4 STATISTICAL ANALYSES

#### 9.4.1 GENERAL APPROACH

Discrete variables will be summarized using frequencies and percentages, while continuous variables will be summarized by means and standard deviations. If the continuous variables are found to be skewed,

we will instead report medians and interquartile ranges. Statistical significance will be determined using p-values less than 0.05 and 95% confidence intervals, unless otherwise indicated. All inferential tests will be two-sided. For descriptive statistics (means, SDs, proportions) where no inferential statistics were conducted, we will refrain from making confirmative statements. All covariates will be pre-specified in the sections below. Any additional analyses will be described as post-hoc and exploratory.

Distribution of the outcome variables will be assessed prior to conduct of our analyses to determine if the planned tests are appropriate. If variables are found to be non-normally distributed we will explore the use of log-transformations or non-parametric tests such as the Wilcoxon-Rank Tests.

# 9.4.2 ANALYSIS OF THE PRIMARY ENDPOINT(S)

The MG-QOL15 scores will be collected for each participant at several time points. The primary outcome, change in MG-QOL15 scores over the first 12-weeks, will be calculated using the first and second collected scores for both groups. Group 1 will have received the full acupuncture intervention between the two measurements while Group 2 will act as the untreated control. We will present the mean change by group with corresponding standard deviations. Analysis of covariances (ANCOVA) with adjustment for baseline MG-QOL15 and covariates identified above will be used to determine if a significant (p<0.05) intervention effect is present. If the model identifies a significant difference in change of MG-QOL15 associated with acupuncture treatment, next steps will assess if this change is still present 12-weeks after completing the full acupuncture treatment. Using data from Group 1, a paired t-test will be used to compare the MG-QOL15 scores directly after treatment (Post-treatment Assessment 1) and scores 12-weeks post-treatment (Post-treatment Assessment 2). (Refer to Schema on page 4 for data collection points.)

Prior to analysis, we will plot our outcomes to examine their distribution and decide whether we should consider non-parametric analyses. Only subjects with complete data from both pre-treatment assessment and 12-week assessment will be included in the final analysis. Data will be analyzed per an intent-to-treat approach regardless of actual treatment received. If a large proportion of missing data is noted, we will compare baseline characteristics of subjects who completed the treatment with those who were lost to follow-up.

# 9.4.3 ANALYSIS OF THE SECONDARY ENDPOINT(S)

Secondary analyses are not dependent on results of primary endpoint. Similar ANCOVA models using data from both groups will be used to determine whether acupuncture treatments were associated with a significant change in MG ADL scores. Before analysis, MG ADL scores will be summarized at each timepoint using measures of center and spread as appropriate.

# 9.4.4 SAFETY ANALYSES

AE/SAEs will be reported as described in **Section 8.3** of this document. They will be classified by severity, relationship to study procedures, and expectedness. No other formal safety analyses will be conducted.

# 9.4.5 BASELINE DESCRIPTIVE STATISTICS

Baseline variables will be compared between groups to ensure randomization achieved balanced treatment assignments. This will include demographics (e.g. gender, age, race). All such variables are

listed in **Section 8.1** of this document. Variables will be summarized using descriptive statistics (e.g. mean and SD, or frequency and proportion) and compared inferentially. Continuous variables will be compared using two-sample t-tests or Wilcoxon rank tests and discrete variables will be compared using chi-square tests for independence or Fisher's exact tests.

#### 9.4.6 PLANNED INTERIM ANALYSES

N/A

#### 9.4.7 SUB-GROUP ANALYSES

Both primary and secondary outcomes will be descriptively summarized based on gender. Our sample size is unlikely to allow for other meaningful sub-group analyses.

#### 9.4.8 TABULATION OF INDIVIDUAL PARTICIPANT DATA

N/A

#### 9.4.9 EXPLORATORY ANALYSES

Exploratory outcomes (medications changes, treatment adherence) will be compared between groups with Student's t-test, Chi-square test, and Mann-Whitney-U test and mixed-model ANOVAs, as appropriate. As an exploratory analysis, patients who report post-COVID-19 symptoms will be identified using the additional COVID-19 set of questions. Types and severity of post-COVID-19 symptoms present within the group will be described. The t-test or non-parametric equivalent will be used to determine whether acupuncture had an effect on post-COVID symptoms.

If necessary, we will conduct a sensitivity analysis in which we exclude participants that had protocol deviations (e.g. large delays between treatments) due to illness, for example COVID-19.

# 10 SUPPORTING DOCUMENTATION AND OPERATIONAL CONSIDERATIONS

# 10.1 REGULATORY, ETHICAL, AND STUDY OVERSIGHT CONSIDERATIONS

# 10.1.1 INFORMED CONSENT PROCESS

# 10.1.1.1 CONSENT/ASSENT AND OTHER INFORMATIONAL DOCUMENTS PROVIDED TO PARTICIPANTS

Consent forms describing in detail the study intervention, study procedures, and risks will be given to the participant and written documentation of informed consent will be completed prior to starting the study intervention. The following consent materials are submitted with this protocol:

- Study Volunteer Informed Consent Form
- Study Participant Informed Consent Form
- Study Participant HIPPA Authorziation Form

- Recruitment Brochure
- Recruitment Flyer

#### 10.1.1.2 CONSENT PROCEDURES AND DOCUMENTATION

At the end of the Pre-screening phone call, all eligible patients will be provided a copy of the consent and HIPPA forms via e-mail. Patients will also be provided an electronic copy of HealthPartners' statement of non-discrimination form. During the Pre-Treatment phone call, research staff will review the consent and HIPAA forms with the patients. Patients will be allowed time to review all documents and ask any questions prior to signing electronically. Research staff will confirm that the patients understand the information in the forms and answer any questions. To obtain signature, the e-consent framework in REDCap will be utilized. This framework allows the patient initials, date, time to be stamped in the footer as extra identity as to who is completing the consent and HIPPA documents. Following the consent conversation, the staff member will sign and e-mail the consent and HIPPA electronically to the patient. The patient will electronically sign, certify, and submit the consent and HIPPA in REDCap. A fully executed PDF copy of the consent and HIPPA will be provided electronically to the patient for their records as well as saved via the auto-archiver function in REDCap. Research staff will complete this process during the Pre-Treatment phone call, to ensure completion and assist if there are any questions.

# 10.1.2 STUDY DISCONTINUATION AND CLOSURE

This study may be temporarily suspended or prematurely terminated if there is sufficient reasonable cause. Written notification, documenting the reason for study suspension or termination, will be provided by the suspending or terminating party to study participants, investigators, the funding agency, the IRB and regulatory authorities. If the study is prematurely terminated or suspended, the PI will promptly inform study participants, the IRB, and the funding agency and will provide the reason(s) for the termination or suspension. Study participants will be contacted, as applicable, and be informed of changes to the study visit schedule.

Circumstances that may warrant termination or suspension include, but are not limited to:

- 1. Determination of unexpected, significant, or unacceptable risk to participants
- 2. Demonstration of efficacy that would warrant stopping
- 3. Insufficient compliance of study staff to the protocol (ie, significant protocol violations)
- 4. Data that are not sufficiently complete and/or evaluable
- 5. Determination of futility

The study may resume once concerns about safety, protocol compliance, and data quality are addressed, and satisfy the funding agency, IRB, or other relevant regulatory or oversight bodies.

#### 10.1.3 CONFIDENTIALITY AND PRIVACY

Participant confidentiality and privacy is strictly held in trust by the participating investigators, their staff, the safety and oversight monitor(s), and the sponsor(s) and funding agency. This confidentiality is extended to the data being collected as part of this study. Data that could be used to identify a specific study participant will be held in strict confidence within the research team. No personally-identifiable information from the study will be released to any unauthorized third party without prior written approval of the sponsor/funding agency.

All research activities will be conducted in as private a setting as possible.

All study regulatory binders will be stored in a locked file cabinet within a secure office. The internal study monitor, representatives of the IRB, or regulatory agencies, may inspect all documents and records required to be maintained by the investigator, for the participants in this study. The clinical study site will permit access to such records.

The study participant's contact information will be securely stored at the clinical site for internal use during the study. At the end of the study, all records will continue to be kept in a secure location for as long a period as dictated by the reviewing IRB, Institutional policies, or sponsor/funding agency requirements.

Study participant research data, which is for purposes of statistical analysis and scientific reporting, will be password-protected and stored on REDCap, a secure web-based system. Only research study staff will have access to the data. Individual participants and their research data will be assigned a unique study identification number. While the study is active, subject identifiers (e.g. name, MRN) will be stored in REDCap, however, after the study is closed all subject identifiers will be removed.

The PI will ensure all mechanisms used to share data will include proper plans and safeguards for the protection of privacy, confidentiality, and security for data dissemination and reuse (e.g., all data will be thoroughly de-identified and will not be traceable to a specific study participant). Plans for archiving and long-term preservation of the data will be implemented, as appropriate.

#### 10.1.4 FUTURE USE OF STORED SPECIMENS AND DATA

After the study is completed, the de-identified data will be and stored in REDCap for use in future research. Permission to keep the de-identified data will be included in the informed consent.

# 10.1.5 KEY ROLES AND STUDY GOVERNANCE

#### **Principal Investigator**

Amanda Herrmann, PhD, Research Associate HealthPartners Neuroscience Center 295 Phalen Blvd. St. Paul, MN 55130 (651) 495-6356 Amanda.A.Herrmann@HealthPartners.com

# 10.1.6 SAFETY OVERSIGHT

There is no Data Safety Monitoring Board for this study, as acupuncture has been previously shown to be safe and have minimal risks. During team meetings, the PI and study will review a rolling report of adverse events and report them appropriately.

#### 10.1.7 CLINICAL MONITORING

N/A, refer to next section.

# 10.1.8 QUALITY ASSURANCE AND QUALITY CONTROL

Study staff will perform internal quality management of study conduct, data collection, documentation and completion.

Quality control (QC) procedures will be implemented as follows:

**Informed consent** --- Study staff will review both the documentation of the consenting process and 10% of the completed consent documents. Feedback will be provided to study staff to ensure proper consenting procedures are followed.

**Source documents and the electronic data ---** The majority of data will be directly entered into eCRFs in REDCap. To ensure accuracy for data not directly entered in REDCap, study staff will compare a representative sample of source data against the database, targeting key data points in that review.

**Intervention Fidelity** — Consistent delivery of the study interventions will be monitored throughout the intervention phase of the study. Procedures for ensuring fidelity of intervention delivery are described in **Section 6.2.1, Interventionist Training and Tracking**.

**Protocol Deviations** – The study team will review documented protocol deviations on an ongoing basis and will implement corrective actions when the quantity or nature of deviations are deemed to be at a level of concern.

We do not anticipate a need for independent monitoring for this study, however, should independent monitoring become necessary, the PI will provide direct access to all trial related sites, source data/documents, and reports for the purpose of monitoring and auditing by the sponsor/funding agency, and inspection by local and regulatory authorities.

#### 10.1.9 DATA HANDLING AND RECORD KEEPING

#### 10.1.9.1 DATA COLLECTION AND MANAGEMENT RESPONSIBILITIES

Data collection will be the responsibility of the research study staff under the supervision of the PI. The PI will be responsible for ensuring the accuracy, completeness, legibility, and timeliness of the data reported.

All data will be entered directly into eCRFs in REDCap. The data system includes password protection and internal quality checks by study staff to identify data that appear inconsistent, incomplete, or inaccurate. Treatment logs from the acupuncture treatment sessions will be scanned into and stored in REDCap.

#### 10.1.9.2 STUDY RECORDS RETENTION

Investigator records will be retained in accordance with regulatory, organizational and sponsor or grantor requirements, but no less than 6 years following the completion of the research. All records will be maintained securely with limited access. Disposal of investigator records will be done in such a manner that no identifying information can be linked to research data.

# 10.1.10 PROTOCOL DEVIATIONS

This protocol defines a protocol deviation as any noncompliance with the clinical trial protocol. The noncompliance may be either on the part of the participant, the investigator, or the study site staff. As a result of deviations, corrective actions will be developed by the site and implemented promptly.

It will be the responsibility of the PI to use continuous vigilance to identify, document, and report deviations as soon as possible, but no later than 10 working days after identification of the protocol deviation. Minor deviations, which do not impact participant safety, compromise the integrity of study data and/or affect the participant's willingness to participate in the research are to be reported at the time of continuing review. Protocol deviations will be addressed in study source documents and sent to the reviewing IRB per their policies. The PI will be responsible for knowing and adhering to the reviewing IRB requirements.

#### 10.1.11 PUBLICATION AND DATA SHARING POLICY

This trial will be registered at ClinicalTrials.gov, and results information from this trial will be submitted to ClinicalTrials.gov. In addition, every attempt will be made to publish results in peer-reviewed journals.

# 10.1.12 CONFLICT OF INTEREST POLICY

The independence of this study from any actual or perceived influence, such as by the pharmaceutical industry, is critical. Therefore, any actual conflict of interest of persons who have a role in the design, conduct, analysis, publication, or any aspect of this trial will be disclosed and managed. Furthermore, persons who have a perceived conflict of interest will be required to have such conflicts managed in a way that is appropriate to their participation in the design and conduct of this trial. The study leadership in conjunction with HealthPartners Institute has established policies and procedures for all study group members to disclose all conflicts of interest and will establish a mechanism for the management of all reported dualities of interest.

# 10.2 ADDITIONAL CONSIDERATIONS

**COVID-19:** This study will align with the HealthPartners' and Park Nicollet's policies regarding COVID-19 for in-person visits. This will be done to ensure the safety of patients and study staff. Appropriate COVID-19 screening procedures and personal protective equipment (PPE) will be utilized for all acupuncture treatment visits. Participants will be screened for COVID-19 on the day of each clinic visit. If a patient screens positive for COVID-19, study visits will be postponed for the appropriate amount of time per current guidance, and we will follow the current clinic site process for COVID-19 positive screens, as defined by the medical group.

#### 10.3 ABBREVIATIONS AND SPECIAL TERMS

| AE | Adverse Event |
|----------------------------|------------------------------|
| ANOVA Analysis of Variance | |
| CFR | Code of Federal Regulations |
| eCRF | Electronic Case Report Forms |
| GCP Good Clinical Practice | |

| HIPPA | Health Insurance Portability and Accountability |
|--------|-------------------------------------------------|
| ICH | International Council on Harmonisation |
| IRB | Institutional Review Board |
| ITT | Intention-To-Treat |
| MG | Myasthenia Gravis |
| OHRP | Office for Human Research Protections |
| PI | Principal Investigator |
| QOL | Quality of Life |
| REDCap | Research Electronic Data Capture |
| SAE | Serious Adverse Event |
| UP | Unanticipated Problem |

# 10.4 PROTOCOL AMENDMENT HISTORY

| Version | Date | Description of Change | Brief Rationale |
|---|---|---|---|
| 2.0 | 01/10/22 | Response to RRC & IRB Review | Addressed reviewer changes |
| 3.0 | 03/02/22 | Removal of electrical stimulation; change inclusion criteria age from 70 to 80; Removal of cardiac/stimulator devices for exclusion as this was specific to electroacupuncture. | Pantheon did not support settings we planned to use and we only planned to stimulate one point. This will not change our hypothesis. Would like to include up to 80 to capture late onset MG. |
| 4.0 | 05/26/22 | Update PN address | Incorrect address |
| 5.0 | 02/16/23 | Add qualitative questions, add letter for recruitment, remove Park Nicollet, and add Como clinic | Adding qualitative survey questions for additional feedback. Sending letter to potentially eligible individuals for recruitment efforts. Removing Park Nicollet clinic and adding Como Clinic for treatment locations. |
| 6.0 | 04/03/23 | Add Stillwater Clinic | Change in locations for acupuncture treatment |
| 7.0 | 09/08/23 | Increase enrollment target to 25. | We are requesting to increase enrollment to 25, so that we can replace any individuals that did not begin treatment. |

# 11 REFERENCES

#### References

- 1. Gilhus NE. Myasthenia Gravis. N Engl J Med. 2016;375(26):2570-2581.
- 2. Carr AS, Cardwell CR, McCarron PO, McConville J. A systematic review of population based epidemiological studies in Myasthenia Gravis. *BMC Neurol.* 2010;10:46.
- 3. Zhang X, Ding W, Wang Z, Gu X, Zhu W. The effectiveness and safety of acupuncture for the treatment of myasthenia gravis: a systematic review and meta-analysis of randomized controlled trials. *Ann Palliat Med.* 2019;8(5):576-585.
- 4. Chon TY, Lee MC. Acupuncture. Mayo Clin Proc. 2013;88(10):1141-1146.
- 5. Yin C, Buchheit TE, Park JJ. Acupuncture for chronic pain: an update and critical overview. *Curr Opin Anaesthesiol.* 2017;30(5):583-592.
- 6. Vickers AJ, Vertosick EA, Lewith G, et al. Acupuncture for Chronic Pain: Update of an Individual Patient Data Meta-Analysis. *J Pain*. 2018;19(5):455-474.
- 7. Chan MWC, Wu XY, Wu JCY, Wong SYS, Chung VCH. Safety of Acupuncture: Overview of Systematic Reviews. *Sci Rep.* 2017;7(1):3369.
- 8. Liu GC, Gao BL, Yang HQ, Qi GY, Liu P. The clinical absolute and relative scoring system-a quantitative scale measuring myasthenia gravis severity and outcome used in the traditional Chinese medicine. *Complement Ther Med.* 2014;22(5):877-886.
- 9. Witt CM, Pach D, Brinkhaus B, et al. Safety of acupuncture: results of a prospective observational study with 229,230 patients and introduction of a medical information and consent form. *Forsch Komplementmed*. 2009;16(2):91-97.
- 10. Hui KK, Nixon EE, Vangel MG, et al. Characterization of the "deqi" response in acupuncture. *BMC Complement Altern Med.* 2007;7:33.
- 11. Lund I, Naslund J, Lundeberg T. Minimal acupuncture is not a valid placebo control in randomised controlled trials of acupuncture: a physiologist's perspective. *Chin Med.* 2009;4:1.
- 12. WHO Standard Acupuncture Point Locations in the Western Pacific Region. World Health Organization, Western Pacific Region; 2008.
- 13. Hoffman JM, Lucas S, Dikmen S, et al. Natural history of headache after traumatic brain injury. *J Neurotrauma*. 2011;28(9):1719-1725.
- 14. Burns TM, Conaway MR, Cutter GR, Sanders DB. Less is more, or almost as much: a 15-item quality-of-life instrument for myasthenia gravis. *Muscle Nerve*. 2008;38(2):957-963.
- 15. Muppidi S. The myasthenia gravis--specific activities of daily living profile. *Ann N Y Acad Sci.* 2012;1274:114-119.